CLINICAL TRIAL: NCT01542983
Title: Feasibility of Prophylactic Treatment of Sleep/Fatigue Before and During Chemotherapy for Breast Cancer
Brief Title: Prophylactic Treatment of Sleep/Fatigue Before and During Chemotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never funded
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sonia Ancoli-Israel, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 120108
Record Dates: First submitted 2012-02-26; First posted 2012-03-02 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Stage, Breast Cancer
Keywords: breast cancer; bright light; insomnia; fatigue
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment-as-usual (Active Comparator): Treatment as usual for fatigue and insomnia
  Interventions: Behavioral: treatment as usual
- Behavioral treatment (Active Comparator): Brief behavioral treatment for insomnia and bright light Light and BBTI combined treatment for insomnia and fatigue
  Interventions: Behavioral: Brief behavioral treatment for insomnia and bright light

INTERVENTIONS:
Behavioral: Brief behavioral treatment for insomnia and bright light — daily bright light exposure; 2 sessions for insomnia
  Arms: Behavioral treatment
Behavioral: treatment as usual — Standard treatment for fatigue and insomnia
  Arms: Treatment-as-usual

SUMMARY:
Women with breast cancer complain of poor sleep and fatigue during chemotherapy which affect their mood, their memory and their quality of life. The investigators are testing whether it is feasible to treat the poor sleep and fatigue with behavioral treatments, before the start of chemotherapy and whether improving sleep and fatigue will also improve mood, memory and quality of life.

DETAILED DESCRIPTION:
Women with breast cancer (BC) report poor sleep and fatigue, occasionally before, and often during chemotherapy. These symptoms often last for months and even years after the end of cancer treatment, significantly burdening the patients' quality of life (QOL), decreasing their overall functional level and potentially hindering the patients' re-integration into productive society. Improvement in the domains of sleep and fatigue might result in overall improvement in QOL. The investigators have shown that women with breast cancer with a symptom cluster of poor sleep, fatigue and depressive symptoms before chemotherapy are more likely to manifest an increase in severity of these symptoms and decreased QOL during chemotherapy.

A randomized controlled treatment study is now warranted to examine whether concurrent treatment of sleep and fatigue, begun before chemotherapy and continuing during chemotherapy, will prevent deterioration of sleep and fatigue during chemotherapy, and since poor sleep and fatigue are related to mood, whether these improvements will then lead to improvements in the symptom cluster of sleep/fatigue/mood as well as in QOL and cognitive functioning during chemotherapy. Before a full study can be initiated, the investigators propose a pilot study to examine the feasibility of conducting this type of treatment study.

The main aims of this pilot study are:

AIM 1: To examine whether the investigators can recruit 20 women with newly diagnosed breast cancer, before they begin chemotherapy, whether or not they are currently experiencing poor sleep and fatigue, into a treatment study that aims at preventing or mitigating poor sleep, fatigue, depressive symptoms during chemotherapy.

AIM 2: To examine whether women recruited into this study will be compliant with the sleep/fatigue treatment for a full four cycles of chemotherapy.

The results of this study plus the preliminary scientific data collected will be used as pilot data for an RO1 with the following aims: Aim 1 - Symptom cluster of sleep/fatigue/mood: To examine the effects of concurrent treatment of poor sleep and fatigue, begun before the start of chemotherapy and continuing during chemotherapy, on the symptom cluster of sleep/fatigue/mood during chemotherapy (hypothesis 1: Women with newly diagnosed breast cancer treated concurrently with Brief Behavioral Treatment of Insomnia (BBTI) and morning bright light therapy (BLT) before the start of and during chemotherapy, will experience fewer symptoms within the cluster of poor sleep, fatigue, depressive symptoms during chemotherapy than women in the information-only control group). Aim 2 - QOL and Cognition: To examine the effects of concurrent treatment of poor sleep and fatigue, begun before the start of chemotherapy and continuing during chemotherapy, on cognitive functioning (as measured with a targeted neuropsychological test battery) and QOL during chemotherapy (hypothesis 2: Women with newly diagnosed breast cancer treated concurrently with BBTI and morning BLT before the start of and during chemotherapy, will experience less deterioration in cognitive functioning and better QOL during chemotherapy than women in the information-only control group).

The innovation of larger application will be that the study intervention is a dual modality intervention (BBTI and BWL), not previously studied in combination and that it ultimately seeks to shift the clinical practice paradigm from a reactive to a proactive, preventive cancer care model.

The investigators are proposing a clinical trial to treat all patients, whether or not they are currently experiencing problems with sleep and fatigue, with the goal of preventing or ameliorating the severity of symptoms during chemotherapy, and compare them to an information-only control group (IC) (see Fig. 1). This pilot study will help us determine the feasibility of such a study.

ELIGIBILITY:
Inclusion Criteria:

* stage I-III breast cancer referred for chemotherapy
* English speaking
* over age 18

Exclusion Criteria:

1. Pregnancy (by self-report; poor sleep and fatigue are sometimes associated with pregnancy);
2. Metastatic or unresectable breast cancer;
3. Patients who have been told they have sleep apnea, restless legs or periodic limb movements in sleep whether or not they are currently treated;
4. History of bipolar disorder or history of mania;
5. Current diagnosis of psychotic disorder;
6. Blindness or other physical or psychological impairments which would limit participation;
7. Shift workers;
8. Women with infants who still disturb the mother's sleep.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
fatigue | 12 weeks
  Change in fatigue from pre-chemotherapy to post cycle 4 chemotherapy

SECONDARY OUTCOMES:
sleep | 12 weeks
  Changes in sleep and sleep quality will be assessed from pre-chemotherapy to post-cycle 4 chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Ancoli-Israel, PhD, Principal Investigator — UCSD
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Study never funded. No data to share